CLINICAL TRIAL: NCT00061854
Title: A Phase II Study Of Intravenous TZT-1027, Administered Weekly Times Two, Every Three Weeks, To Patients With Progressive Locally Advanced Or Metastatic Non-Small Cell Lung Cancer (NSCLC) Following Treatment With Platinum-Based Chemotherapy
Brief Title: Soblidotin in Treating Patients With Progressive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000301749; DAIICHI-1027A-PRT005; MSKCC-03016
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — soblidotin

INTERVENTIONS:
Drug: soblidotin

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as soblidotin use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of soblidotin in treating patients who have progressive locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate and duration of response in patients with progressive locally advanced or metastatic non-small cell lung cancer treated with soblidotin as second-line therapy after receiving prior platinum-based chemotherapy.
* Determine the time to tumor progression in patients treated with this drug.
* Determine the median survival time and 12-month survival rate of patients treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive soblidotin IV over 1 hour on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Plasma sampling for pharmacokinetics is done on day 1 of course 1.

Patients are followed for survival every 3 months after discontinuing study treatment.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Locally advanced or metastatic disease
* Demonstrates tumor progression
* Must have received 1 prior chemotherapy regimen

  * Prior chemotherapy must have included a platinum agent
* Measurable disease

  * At least 1 measurable lesion outside the field of any prior radiotherapy
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiac

* Ejection fraction at least 40% by MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric disorder that would preclude giving informed consent or following study instruction
* No grade 2 or greater neurotoxicity
* No other prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix unless in complete remission and off therapy for that disease for at least 5 years prior to study entry
* No other concurrent severe or uncontrolled underlying medical disease that would compromise patient safety and study outcome
* No concurrent serious infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No concurrent anticancer radiotherapy

  * Concurrent localized radiotherapy to a non-indicator lesion for pain relief is allowed provided other methods of pain control are ineffective

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* At least 4 weeks since prior myelosuppressive therapy
* More than 28 days since prior investigational drugs
* No other concurrent investigational drugs
* No other concurrent anticancer cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cheverton, MD, ChB, MMED, RadT, Study Chair — Daiichi Pharmaceuticals
Locations (3):
- United States (3):
  - Medical Oncology and Hematology, P.C., Waterbury, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York